CLINICAL TRIAL: NCT01501448
Title: Oral Estradiol Valerate Versus Oral Contraceptive Pill in Invitro Fertilization Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: IVI Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IVIMAD-GV-OCPE-2011
Record Dates: First submitted 2011-12-27; First posted 2011-12-29 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Ethinyl Estradiol-Norgestrel Combination; Estradiol

ARMS (2):
- OCP (Active Comparator)
  Interventions: Drug: Levonorgestrel and ethinylestradiol
- Oral estradiol valerate (Active Comparator)
  Interventions: Drug: Estradiol valerate

INTERVENTIONS:
Drug: Levonorgestrel and ethinylestradiol — 30 microgram of ethinylestradiol plus levonorgestrel daily for 12 to 16 days
  Arms: OCP
Drug: Estradiol valerate — 4mg estradiol valerate from cycle day 20 till the day before the initiation of the cycle
  Arms: Oral estradiol valerate

SUMMARY:
The recent controversy regarding the use of pill for cycle planning in GnRH antagonists IVF cycle has driven the search for new ways to plan IVF cycles in order to avoid weekends or to equally distribute the workload. Recently, mid-late luteal phase oral estrogens seem to be as good as the pill. The investigators will compare OCP vs oral estrogens to plan the initiation of IVF cycles.

ELIGIBILITY:
Inclusion Criteria:

* 1st or 2nd IVF cycle
* BMI <30 kg/m2
* regular menstrual cycles
* basal FSH <10IU and E2 <60pg/mL

Exclusion Criteria:

* polycystic ovaries
* endometriosis
* previous ovarian surgery
* previous low ovarian response

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Implantation rate | 20 days after the embryo transfer
  number of embryonic sacs visible by ultrasound divided by the number of embryos transferred

CONTACTS AND LOCATIONS:
Locations (1):
- IVI Madrid, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Hauzman EE, Zapata A, Bermejo A, Iglesias C, Pellicer A, Garcia-Velasco JA. Cycle scheduling for in vitro fertilization with oral contraceptive pills versus oral estradiol valerate: a randomized, controlled trial. Reprod Biol Endocrinol. 2013 Sep 28;11:96. doi: 10.1186/1477-7827-11-96. PMID 24074027